CLINICAL TRIAL: NCT05467293
Title: A Phase 2, Multi-center, Randomized, Double- Masked and Placebo-Controlled Study Evaluating the Efficacy and Safety of YP-P10 Ophthalmic Solution Compared to Placebo in Subjects With Dry Eye (ICECAP 1)
Brief Title: Phase 2, Multi-center, Randomized, Double- Masked and Placebo-Controlled Study of YP-P10 Ophthalmic Solution Compared to Placebo in Subjects With Dry Eye (ICECAP 1)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yuyu Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YPP10-001
Record Dates: First submitted 2022-06-28; First posted 2022-07-20 (Actual); Results first posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: multicenter, randomized, double-masked, placebo-controlled clinical study. Subjects will be randomized to one of the following treatment arms at Visit 2 (Day 1):
  * 0.3% YP-P10 Ophthalmic Solution: 1 drop BID in each eye (N = ~80)
  * 1% YP-P10 Ophthalmic Solution: 1 drop BID in each eye (N = ~80)
  * YP-P10 Placebo Ophthalmic Solution (vehicle): 1 drop BID in each eye (N = ~80)
Who Masked: Participant, Care Provider, Investigator
Masking Description: Before the initiation of study run-in at Visit 1, each subject who provides written informed consent will be assigned a screening number. All screening numbers will be assigned in strict numerical sequence at a site and no numbers will skipped or omitted. Each subject who meets all the inclusion and none of the exclusion criteria at Visit 1 and Visit 2 will be assigned a randomization number at the end of Visit 2. The Interactive Web Response System (IWRS) will be used to assign all randomization numbers.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 0.3% YP-P10 Ophthalmic Solution (Active Comparator)
  Interventions: Drug: 0.3% YP-P10 Ophthalmic Solution
- 1% YP-P10 Ophthalmic Solution (Active Comparator)
  Interventions: Drug: 1% YP-P10 Ophthalmic Solution
- YP-P10 Placebo Ophthalmic Solution (vehicle) (Placebo Comparator)
  Interventions: Drug: YP-P10 Placebo Ophthalmic Solution (vehicle)

INTERVENTIONS:
Drug: 0.3% YP-P10 Ophthalmic Solution — Drug: YP-P10 Ophthalmic Solution
  Arms: 0.3% YP-P10 Ophthalmic Solution
Drug: 1% YP-P10 Ophthalmic Solution — Drug: YP-P10 Ophthalmic Solution
  Arms: 1% YP-P10 Ophthalmic Solution
Drug: YP-P10 Placebo Ophthalmic Solution (vehicle) — Placebo YP-P10 Placebo Ophthalmic Solution (vehicle)
  Arms: YP-P10 Placebo Ophthalmic Solution (vehicle)

SUMMARY:
The objective of this study is to compare the safety and efficacy of YP-P10 Ophthalmic Solution to placebo for the treatment of the signs and symptoms of dry eye.

DETAILED DESCRIPTION:
The clinical hypotheses for this study is that 0.3% YP-P10 Ophthalmic Solution twice daily (BID) and 1.0% YP-P10 Ophthalmic Solution BID are superior to YP-P10 Placebo Ophthalmic Solution (vehicle) for the primary endpoints of signs and symptoms of dry eye, as follows:

* Sign: Total corneal fluorescein staining score of the study eye using the modified NEI grading scale, measured by mean change from baseline (Visit 2, Pre- Controlled Adverse Environment [CAE®]) to Visit 6
* Symptom: Ocular discomfort score of both eyes using the Visual Analog Scale (VAS) Ocular Discomfort Scale, measured by mean change from baseline (Visit 2, Pre-CAE®) to Visit 6

ELIGIBILITY:
Inclusion Criteria:

• Individuals eligible to participate in this study must meet all of the following criteria: 0. Be at least 18 years of age;

1. Provide written informed consent;
2. Be willing and able to comply with all study procedures;
3. Have a patient-reported history of dry eye for at least 6 months prior to Visit 1;
4. Have a history of use or desire to use eye drops for dry eye symptoms within 6 months of Visit 1;
5. Have a best corrected visual acuity (BCVA) of 0.7 logarithm of the minimum angle of resolution (logMAR) or better (Snellen equivalent score of 20/100 or better) in each eye at Visit 1;
6. Have a score of ≥ 2 for both eyes according to the Ora Calibra® Ocular Discomfort & 4- Symptom Questionnaire in at least one of the dry eye symptoms at Visits 1 and 2;
7. Have an unanesthetized Schirmer's Test score of ≤ 10 mm/5 minutes and ≥ 1 mm/5 minutes in at least one eye at Visits 1 and 2;
8. Have a corneal fluorescein staining score of ≥ 2 according to the Ora Calibra® Corneal and Conjunctival Staining Scale for Grading of Fluorescein Staining in at least one region in one eye at Visits 1 and 2 and a central score ≥ 1 in the same eye;
9. Have a conjunctival redness score ≥ 1 according to the Ora Calibra® Conjunctival Redness for Dry Eye Scale in at least one eye at Visits 1 and 2 pre-CAE®;
10. Demonstrate in the same eye(s) a response to the CAE® at Visits 1 and 2 as defined by:

    * Having at least a ≥1 point increase in fluorescein staining in the inferior region in at least one eye following CAE® exposure; a. Reporting an Ocular Discomfort score ≥ 3 at 2 or more consecutive time points in at least one eye during CAE® exposure (if a subject has an Ocular Discomfort rating of 3 at time = 0 for an eye, s/he must report an Ocular Discomfort rating of 4 for two consecutive measurements for that eye). Note: a subject cannot have an Ocular Discomfort score of 4 at time = 0);
11. Have at least one eye, the same eye, satisfy all criteria for 8, 9, 10 and 11 above;
12. A negative urine pregnancy test if female of childbearing potential (those who are not surgically sterilized [bilateral tubal ligation, hysterectomy or bilateral oophorectomy] or post-menopausal [12 months after last menses]) and must use adequate birth control through the study period. For non-sexually active females, abstinence may be regarded as an adequate method of birth control.)

Exclusion Criteria:

• Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study: 0. Have any clinically significant slit lamp findings at Visit 1 that may include active blepharitis, meibomian gland dysfunction, lid margin inflammation, or active ocular allergies that require therapeutic treatment, and/or in the opinion of the investigator may interfere with study parameters;

1. Be diagnosed with an ongoing ocular infection (bacterial, viral, or fungal), or active ocular inflammation at Visit 1;
2. Have worn contact lenses within 7 days of Visit 1 or anticipate using contact lenses during the study;
3. Have previously had laser-assisted in situ keratomileusis (LASIK) surgery within the last 12 months;
4. Have used Restasis®, Xiidra®, or Cequa®, Eysuvis™ and Tyrvaya™ within 60 days of Visit 1;
5. Have had any ocular and/or lid surgeries in the past 6 months or have any planned ocular and/or lid surgeries over the study period;
6. Be using or anticipate using temporary punctal plugs during the study that have not been stable within 30 days of Visit 1;
7. Be currently taking any topical ophthalmic prescription (including medications for glaucoma) or over-the-counter solutions, artificial tears, gels or scrubs, and cannot discontinue these medications for the duration of the trial (excluding medications allowed for the conduct of the study); the respective wash- out periods are required for the following medications:

   * Antihistamines (including ocular): 72 hours prior to Visit 1

     1. Oral aspirin or aspirin-containing products allowed if dose has been stable over past 30 days prior to Visit 1 and no change in dose is anticipated during the study period
     2. Corticosteroids or mast cell stabilizers (including ocular): 14 days prior to Visit 1
     3. Any medication (oral or topical) known to cause ocular drying that has not been administered as a stable dose for at least 30 days prior to Visit 1 and during the study
     4. All other topical ophthalmic preparations (including artificial tear substitutes) other than the study drops: 72 hours prior to Visit 1
8. Have an uncontrolled systemic disease;
9. Be a woman who is pregnant, nursing, or planning a pregnancy;
10. Be unwilling to submit a urine pregnancy test at Visit 1 and Visit 6 (or early termination visit) if of childbearing potential. Non- childbearing potential is defined as a woman who is permanently sterilized (e.g., has had a hysterectomy or tubal ligation), or is post- menopausal (without menses for 12 consecutive months);
11. Be a woman of childbearing potential who is not using an acceptable means of birth control; acceptable methods of contraception include: hormonal - oral, implantable, injectable, or transdermal contraceptives; mechanical - spermicide in conjunction with a barrier such as a diaphragm or condom; intrauterine device; or surgical sterilization of partner. For non-sexually active females, abstinence may be regarded as an adequate method of birth control; however, if the subject becomes sexually active during the study, she must agree to use adequate birth control as defined above for the remainder of the study;
12. Have a known allergy and/or sensitivity to the test article or its components;
13. Have a condition or be in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study;
14. Be currently enrolled in an investigational drug or device study or have used an investigational drug or device within 30 days of Visit 1;
15. Be unable or unwilling to follow instructions, including participation in all study assessments and visits.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-03-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Cornea Consultants of Arizona, Phoenix, Arizona
  - Aesthetic Eye Care Institute, Newport Beach, California
  - Vision Institute, Colorado Springs, Colorado
  - Andover Eye Associates, Andover, Massachusetts
  - NC Eye Associates, Apex, North Carolina
  - Oculus Research, Garner, North Carolina
  - Total Eye Care, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.3% YP-P10 Ophthalmic Solution: Participants enrolled in 0.3% YP-P10 Ophthalmic Solution: Drug: YP-P10 Ophthalmic Solution group
- 1% YP-P10 Ophthalmic Solution: Participants enrolled in 1% YP-P10 Ophthalmic Solution: Drug: YP-P10 Ophthalmic Solution group
- YP-P10 Placebo Ophthalmic Solution (Vehicle): Participants enrolled in YP-P10 Placebo Ophthalmic Solution (vehicle): Placebo YP-P10 Placebo Ophthalmic Solution (vehicle) group
Period: Overall Study
Arm/Group | 0.3% YP-P10 Ophthalmic Solution | 1% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Started | 85 | 86 | 86
Completed | 77 | 81 | 84
Not Completed | 8 | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.3% YP-P10 Ophthalmic Solution | 1% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle) | Total
Number analyzed (Participants) | 85 | 86 | 86 | 257
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | NA — Participants must be over 18 years old to partake in study | NA — Participants must be over 18 years old to partake in study | NA — Participants must be over 18 years old to partake in study | NA — Total not calculated because data are not available (NA) in one or more arms.
  Between 18 and 65 years | 46 | 51 | 48 | 145
  >=65 years | 39 | 35 | 38 | 112
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 59 | 61 | 192
  Male | 13 | 27 | 25 | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 1 | 3
  Asian | 16 | 17 | 17 | 50
  Black or African American | 23 | 17 | 14 | 54
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  White | 44 | 50 | 52 | 146
  Other | 0 | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 85 | 86 | 86 | 257
Ethnicity [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 9 | 11 | 33
  Not Hispanic or Latino | 72 | 77 | 75 | 224
Iris Color (OD) [Count of Participants; unit: Participants]
  Black | 3 | 2 | 2 | 7
  Blue | 8 | 13 | 11 | 32
  Brown | 59 | 55 | 54 | 168
  Hazel | 8 | 8 | 10 | 26
  Green | 7 | 8 | 9 | 24
  Gray | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0
Iris Color (OS) [Count of Participants; unit: Participants]
  Black | 3 | 2 | 2 | 7
  Blue | 8 | 13 | 11 | 32
  Brown | 59 | 55 | 54 | 168
  Hazel | 8 | 8 | 10 | 26
  Green | 7 | 8 | 9 | 24
  Gray | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Total Corneal Fluorescein Staining
Description: Modified National Eye Institute Scale; 0-20: Higher is Worse
Time Frame: Day 85
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Number analyzed (Eyes) | 172 | 170 | 172
score on a scale | 7.35 (1.730) | 7.25 (1.957) | 7.12 (1.850)

2. Primary Outcome: Ocular Discomfort Score
Description: Visual Analogue Scale; 0-100: Higher is Worse
Time Frame: Day 85
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Number analyzed (Eyes) | 172 | 170 | 172
score on a scale | 52.8 (24.77) | 54.2 (27.17) | 53.6 (26.40)

3. Secondary Outcome: Fluorescein Staining: Inferior
Description: Modified National Eye Institute Scale; 0-4: Higher is Worse
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Number analyzed (Eyes) | 172 | 170 | 172
score on a scale | 1.71 (0.379) | 1.71 (0.471) | 1.73 (0.507)

4. Secondary Outcome: Fluorescein Staining: Superior
Description: Modified National Eye Institute Scale; 0-4: Higher is Worse
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Number analyzed (Eyes) | 172 | 170 | 172
score on a scale | 1.34 (0.516) | 1.36 (0.537) | 1.26 (0.519)

5. Secondary Outcome: Fluorescein Staining: Central
Description: Modified National Eye Institute Scale; 0-4: Higher is Worse
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Number analyzed (Eyes) | 172 | 170 | 172
score on a scale | 1.33 (0.535) | 1.28 (0.543) | 1.29 (0.545)

6. Secondary Outcome: Fluorescein Staining: Temporal
Description: Modified National Eye Institute Scale; 0-4: Higher is Worse
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Number analyzed (Eyes) | 172 | 170 | 172
score on a scale | 1.36 (0.501) | 1.33 (0.570) | 1.29 (0.444)

7. Secondary Outcome: Fluorescein Staining: Nasal
Description: Modified National Eye Institute Scale; 0-4: Higher is Worse
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Number analyzed (Eyes) | 172 | 170 | 172
score on a scale | 1.60 (0.548) | 1.57 (0.655) | 1.55 (0.542)

8. Secondary Outcome: Lissamine Green Staining: Conjunctival Sum
Description: Modified National Eye Institute Scale; 0-24: Higher is Worse
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Number analyzed (Eyes) | 172 | 170 | 172
score on a scale | 5.36 (3.922) | 4.96 (3.872) | 5.62 (3.848)

9. Secondary Outcome: Lissamine Green Staining: Inferior Temporal
Description: Modified National Eye Institute Scale; 0-4: Higher is Worse
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Number analyzed (Eyes) | 172 | 170 | 172
score on a scale | 0.83 (0.754) | 0.76 (0.680) | 0.95 (0.695)

10. Secondary Outcome: Lissamine Green Staining: Superior Temporal
Description: Modified National Eye Institute Scale; 0-4 Higher is Worse
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Number analyzed (Eyes) | 172 | 170 | 172
score on a scale | 0.76 (0.689) | 0.66 (0.700) | 0.76 (0.723)

11. Secondary Outcome: Lissamine Green Staining: Temporal
Description: Modified National Eye Institute Scale; 0-4 Higher is Worse
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Number analyzed (Eyes) | 172 | 170 | 172
score on a scale | 0.88 (0.747) | 0.81 (0.802) | 0.93 (0.760)

12. Secondary Outcome: Lissamine Green Staining: Inferior Nasal
Description: Modified National Eye Institute Scale; 0-4 Higher is Worse
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Number analyzed (Eyes) | 172 | 170 | 172
score on a scale | 0.92 (0.751) | 0.94 (0.775) | 1.11 (0.733)

13. Secondary Outcome: Lissamine Green Staining: Superior Nasal
Description: Modified National Eye Institute Scale; 0-4 Higher is Worse
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Number analyzed (Eyes) | 172 | 170 | 172
score on a scale | 0.94 (0.799) | 0.86 (0.830) | 0.88 (0.818)

14. Secondary Outcome: Lissamine Green Staining: Nasal
Description: Modified National Eye Institute Scale; 0-4 Higher is Worse
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Number analyzed (Eyes) | 172 | 170 | 172
score on a scale | 1.04 (0.862) | 0.93 (0.810) | 0.99 (0.799)

15. Secondary Outcome: Conjunctival Redness
Description: Ora Calibra Scale; 0-4 Higher is Worse
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Number analyzed (Eyes) | 172 | 170 | 172
score on a scale | 1.87 (0.619) | 1.87 (0.655) | 1.94 (0.639)

16. Secondary Outcome: Unanesthetized Schirmer's Test
Description: score on a scale of ≤ 10 mm/5 minutes and ≥ 1 mm/5 minutes in at least one eye. Schirmer's test can be interpreted as follows: 0 to 5 mm: extremely dry eyes; 5 to 10 mm: moderately dry eyes; 10 to 15 mm: possible dry eyes; Longer than 15 mm: normal tear function.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Eyes
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Number analyzed (Eyes) | 172 | 170 | 172
mm | 5.2 (2.82) | 5.0 (2.76) | 4.7 (2.72)

17. Secondary Outcome: Tear Film Break-up Time (TFBUT)
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: Eyes
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Number analyzed (Eyes) | 172 | 170 | 172
seconds | 2.598 (0.8443) | 2.540 (0.9201) | 2.441 (0.8812)

18. Secondary Outcome: Ocular Surface Disease Index (OSDI): Subtotal 1-5
Description: Ocular Surface Disease Index Scale 0-100 (higher is worse)
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Number analyzed (Eyes) | 172 | 170 | 172
score on a scale | 37.44 (19.804) | 37.71 (21.555) | 37.50 (17.485)

19. Secondary Outcome: Ocular Surface Disease Index (OSDI): Subtotal 6-9
Description: Ocular Surface Disease Index Scale 0-100 (higher is worse)
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Number analyzed (Eyes) | 172 | 170 | 172
score on a scale | 39.29 (24.653) | 40.34 (27.580) | 35.75 (22.152)

20. Secondary Outcome: Ocular Surface Disease Index (OSDI): Subtotal 10-12
Description: Ocular Surface Disease Index Scale 0-100 (higher is worse)
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Number analyzed (Eyes) | 172 | 170 | 172
score on a scale | 55.86 (27.538) | 49.26 (27.346) | 55.53 (26.114)

21. Secondary Outcome: Ocular Surface Disease Index (OSDI): Total
Description: Ocular Surface Disease Index Scale 0-100 (higher is worse)
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Number analyzed (Eyes) | 172 | 170 | 172
score on a scale | 42.49 (19.426) | 41.46 (20.031) | 41.42 (17.098)

22. Secondary Outcome: Burning/Stinging
Description: Visual Analog Scale; 0-100: Higher is Worse
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Number analyzed (Eyes) | 172 | 170 | 172
score on a scale | 34.5 (25.56) | 37.9 (28.33) | 43.3 (26.48)

23. Secondary Outcome: Itching
Description: Visual Analog Scale; 0-100: Higher is Worse
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Number analyzed (Eyes) | 172 | 170 | 172
score on a scale | 38.5 (25.05) | 44.2 (28.09) | 40.9 (25.50)

24. Secondary Outcome: Foreign Body Sensation
Description: Visual Analog Scale; 0-100: Higher is Worse
Time Frame: 13 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Number analyzed (Eyes) | 172 | 170 | 172
score on a scale | 38.8 (27.62) | 40.2 (28.63) | 40.6 (28.46)

25. Secondary Outcome: Blurred Vision
Description: Visual Analog Scale; 0-100: Higher is Worse
Time Frame: 13 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Number analyzed (Eyes) | 172 | 170 | 172
score on a scale | 41.2 (27.90) | 45.0 (28.89) | 41.5 (26.62)

26. Secondary Outcome: Eye Dryness
Description: Visual Analog Scale; 0-100: Higher is Worse
Time Frame: 13 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Number analyzed (Eyes) | 172 | 170 | 172
score on a scale | 61.2 (24.50) | 65.3 (23.51) | 60.4 (23.42)

27. Secondary Outcome: Photophobia
Description: Visual Analog Scale; 0-100: Higher is Worse
Time Frame: 13 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Number analyzed (Eyes) | 172 | 170 | 172
score on a scale | 44.9 (27.70) | 47.1 (29.82) | 44.0 (29.57)

28. Secondary Outcome: Pain in Eyes
Description: Visual Analog Scale; 0-100: Higher is Worse
Time Frame: 13 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Number analyzed (Eyes) | 172 | 170 | 172
score on a scale | 30.5 (27.26) | 28.2 (25.64) | 33.6 (28.10)

29. Secondary Outcome: Treatment Compliance Using a Daily Compliance Diary
Description: Self-Administrating with use of Daily Compliance Diary. Subject daily diaries were collected at Visits 1 through 6, and the subject's used and unused study drug ampules were collected at Visit 3 through 6. Dosing compliance was based on the used and unused ampule count. If the subject was less than 80% or more than 125% compliant with dosing based on the expected number of used ampules, then the subject was deemed noncompliant and a dosing deviation was recorded.
  Dosing compliance (% compliance) was assessed by calculating the number of actual doses received and comparing that to the number of expected doses as follows:
  Compliance (%) = Number of Actual Doses Received / Number of Expected Doses x 100%
  The number of expected doses that will be used for calculating compliance was calculated as:
  2 x [(Date of Last Dose - Date of First Dose) + 1]
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: percentage of compliance
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
percentage of compliance | 114.90 (134.816) | 100.13 (4.525) | 100.83 (8.480)

30. Secondary Outcome: Drop Comfort - Positive Response
Description: A drop comfort evaluation will be performed immediately upon administration of study drug and then at 1, 2, and 3 minutes following initial dosing using the Ora Calibra Drop Comfort Scale
Time Frame: 13 weeks
Measure: Median (Full Range); unit: percentage of comfort
Units Other Than Participants: Eyes
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Number analyzed (Eyes) | 172 | 170 | 172
percentage of comfort | 89.5 [0 to 100] | 84.7 [0 to 100] | 84.9 [0 to 100]

31. Secondary Outcome: Visual Acuity - Subjects With Increase Greater Than 0.2 logMAR
Description: Visual Acuity was assessed using an ETDRS chart
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Participants | 0 | 0 | 0

32. Secondary Outcome: Slit-lamp Evaluation Biomicroscopy - Subjects That Had a Shift From Normal/Abnormal NCS to Abnormal CS
Description: Slit lamp biomicroscopic observations will be graded as Normal or Abnormal
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Participants | 0 | 0 | 0

33. Secondary Outcome: Adverse Event Query - TEAEs
Description: Each subject will be queried regarding adverse events
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Participants | 21 | 24 | 31

34. Secondary Outcome: Adverse Event Query - Ocular TEAEs
Description: Each subject will be queried regarding adverse events
Time Frame: 13 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Participants | 12 | 13 | 17

35. Secondary Outcome: Adverse Event Query - Non Ocular TEAEs
Description: Each subject will be queried regarding adverse events
Time Frame: 13 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Participants | 11 | 13 | 18

36. Secondary Outcome: Adverse Event Query - TEAEs Causing Premature Treatment Discontinuation
Description: Each subject will be queried regarding adverse events
Time Frame: 13 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Participants | 3 | 2 | 1

37. Secondary Outcome: Adverse Event Query - TEAEs Suspected to be Related to Study Drug
Description: Each subject will be queried regarding adverse events
Time Frame: 13 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Participants
  Definitely related to study drug | 8 | 5 | 5
  Probably related to study drug | 2 | 1 | 4
  Possibly related to study drug | 1 | 2 | 4
  No TEAE Reported | 75 | 77 | 73

38. Secondary Outcome: Adverse Event Query - SEA Reported
Description: Each subject will be queried regarding adverse events
Time Frame: 13 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Participants | 1 | 0 | 1

39. Secondary Outcome: Dilated Fundoscopy: Shift From Normal/Abnormal NCS to Abnormal CS
Description: using indirect ophthalmoscopy. The Investigator will make observations of the vitreous, retina, macula, choroid and optic nerve.
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Participants | 0 | 0 | 0

40. Secondary Outcome: Intraocular Pressure (IOP) by Contact Tonometry by the Examiner: Unsafe and Abnormal Ranges
Description: A single measurement is made
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 86 | 85 | 86
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 13 Weeks
Arm/Group | 1% YP-P10 Ophthalmic Solution | 0.3% YP-P10 Ophthalmic Solution | YP-P10 Placebo Ophthalmic Solution (Vehicle)
All-Cause Mortality (participants affected / at risk) | 1/86 | 0/85 | 0/86
Serious Adverse Events (participants affected / at risk) | 1/86 | 0/85 | 1/86
Other Adverse Events (participants affected / at risk) | 28/86 | 34/85 | 42/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1% YP-P10 Ophthalmic Solution (N=86) | 0.3% YP-P10 Ophthalmic Solution (N=85) | YP-P10 Placebo Ophthalmic Solution (Vehicle) (N=86)
Serious Adverse Event (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Cardiac arrest secondary to arteriosclerotic cardiovascular disease leading to death
Serious Adverse Event (General disorders) | 0 (0) | 0 (0) | 1 (1) — Worsening of laceration in the right leg
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1% YP-P10 Ophthalmic Solution (N=86) | 0.3% YP-P10 Ophthalmic Solution (N=85) | YP-P10 Placebo Ophthalmic Solution (Vehicle) (N=86)
Instillation Eye Pain (General disorders) | 10 (10) | 4 (4) | 9 (9)
Visual acuity reduced (Eye disorders) | 1 (1) | 3 (3) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 2 (2)
Acquired hypertrophy of the retinal pigment epithelium (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Blindness (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Corneal infiltrates (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eyelid myokymia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Foreign body sensation in eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Ocular discomfort (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Visual Impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Conjunctival abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 2 (2) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Contision (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ligament Sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Greater trochanteric pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intravertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic, and mediastinal disorders (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Oropharyngeal pain (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Keloid scar (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/93/NCT05467293/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-09): https://cdn.clinicaltrials.gov/large-docs/93/NCT05467293/SAP_001.pdf